CLINICAL TRIAL: NCT01208285
Title: A Phase 1 Non-Randomized, Open-Label Study to Assess the Safety and Pharmacokinetics of VX-770 in Subjects With Moderate Hepatic Impairment and in Matched Healthy Subjects
Brief Title: Study of VX-770 in Subjects With Moderate Hepatic Impairment and in Matched Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Medical Monitor, Vertex Pharmaceuticals Incorporated
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX10-770-013
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: In Development for Cystic Fibrosis
MeSH Terms: interventions — ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): approximately 12 male and female subjects with moderate hepatic impairment
  Interventions: Drug: VX-770
- Group B (Experimental): approximately 12 healthy male and female subjects
  Interventions: Drug: VX-770

INTERVENTIONS:
Drug: VX-770 — 150 mg oral tablet

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics and safety of a single dose of VX-770 in subjects with moderate hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

Group A (Subjects with Hepatic Impairment):

* male or female between 18 and 65 years of age
* subjects must have a Child-Pugh total score of 7 to 9
* subjects must agree to use 1 highly effective method of contraception during the study and for 90 days after the completion of the study
* subjects must have a body mass index (BMI) of 18 to 35 kg/m2

Group B (Healthy Subjects):

* male or female between 18 and 65 years of age
* subjects will match subjects with hepatic impairment for sex, BMI, cigarette smoking habit, and age
* subjects must agree to use 1 highly effective method of contraception during the study and for 90 days after the completion of the study

Exclusion Criteria:

Group A (Subjects with Hepatic Impairment):

* subjects who are not clinically stable or who have a history of any illness that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject
* subjects who are unwilling or unable to discontinue use of any inhibitors or inducers of CYP3A
* subjects who have a history of alcohol abuse within 1 year or illicit drug abuse within 2 years
* subjects who smoke more than 10 cigarettes per day
* subjects who have fluctuating or rapidly deteriorating hepatic function
* subjects who have significant renal dysfunction
* subjects who have HIV, or active hepatitis B
* subjects who have previous solid organ or bone marrow transplantation

Group B (Healthy Subjects):

* subjects who have a history of any illness that, in the opinion of the investigator or the subject's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the subject
* subjects who are unwilling or unable to discontinue use of any inhibitors or inducers of CYP3A
* subjects who have a history of alcohol or illicit drug abuse within 2 years
* subjects who smoke more than 10 cigarettes per day
* subjects who have HIV, hepatitis C, or active hepatitis B

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
VX-770 pharmacokinetic parameters | 4 or 10 Days

SECONDARY OUTCOMES:
VX-770 metabolites pharmacokinetic parameters | 4 or 10 days
Safety as measured by adverse events, clinical laboratory values, standard electrocardiograms (ECGs), and vital signs | up to 40 days

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (2):
  - Hradec Králové
  - Prague
- Bratislava, Slovakia